CLINICAL TRIAL: NCT02619838
Title: Prospective Subtalar, Double, or Triple Arthrodesis Study With CCS Screws
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Medartis AG (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro00059296
Record Dates: First submitted 2015-10-15; First posted 2015-12-02 (Estimated); Results first posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Post-traumatic Osteoarthritis, Unspecified Ankle and Foot; Localized, Primary Osteoarthritis of the Ankle and/or Foot
Keywords: Double Arthrodesis; Triple Arthrodesis; Subtalar Arthrodesis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Aptus CCS 5.0 or/and 7.0 screws: Procedure/Surgery: Subtalar, Double or Triple Arthrodesis of the talonavicular joint, the subtalar joint, and the calcaneal-cuboid joint of the foot with the Aptus CCS 5.0 or/and 7.0 screws
  Interventions: Device: Aptus CCS 5.0 or/and 7.0 screws

INTERVENTIONS:
Device: Aptus CCS 5.0 or/and 7.0 screws — Fusion of the talonavicular joint, the subtalar joint, and the calcaneal-cuboid joint with a Aptus CCS screws. The assignment of the device is at the discretion of the standard of care provider, not the study investigator.

SUMMARY:
The objective of this study is to prospectively evaluate the mid-term results and intraoperative and postoperative complication rate in patients who underwent double or triple arthrodesis using CCS screws.

DETAILED DESCRIPTION:
This proposal is a collaborative effort of Medartis. This is a prospective investigation to evaluate the mid-term results and intraoperative and postoperative complication rate in patients who underwent subtalar,double or triple arthrodesis using CCS screws.The assignment of the device is at the discretion of the standard of care provider, not the study investigator.

Patients undergoing a double or triple arthrodesis in their foot using Aptus CCS screws will be asked to enroll in this study. After informed consent, the patients will be asked to complete the following patient reported outcomes questionnaires (standard of care for all patients in the Foot and Ankle section): VAS for pain, modified Coughlin rating scale, AOFAS, and FADI at each standard of care visit which includes preoperative, 6 weeks, 3 months, 6 months, 1 year, and 2 years post operative. Patients will also receive standard of care radiographs at these visits, and a standard of care CT scan at 6 months.

Patients will be identified in the clinic by an attending orthopaedic foot and ankle surgeon or his physician assistant based on clinical exam and radiographic findings. Inclusion criteria include anyone over age 18 who has Rheumatoid or posttraumatic osteoarthritis of the hindfoot with involvement of subtalar, talonavicular, and calcaneocuboid joints, and/or Symptomatic rigid pes planovalgus et abductus with end-stage posterior tibial tendon dysfunction, and/or Neuromuscular disease mediated hindfoot deformities, and/or Tarsal coalitions, and/or Indication for calcaneocuboid arthrodesis: severe degenerative changes in the calcaneocuboid joint and/or severe abductus deformity of the forefoot.and has failed nonoperative management. Typically, these patients have multiple medical comorbidities and therefore the only exclusion criteria will be patients who are not healthy enough to undergo surgery. Approximately 50 patients will be recruited for the study.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid or posttraumatic osteoarthritis of the hindfoot with involvement of subtalar, talonavicular, and calcaneocuboid joints (2;12).
* Symptomatic rigid pes planovalgus et abductus with end-stage posterior tibial tendon dysfunction (e.g. grade IV) (4;13-15).
* Neuromuscular disease mediated hindfoot deformities (16).
* Tarsal coalitions (17).
* Indication for calcaneocuboid arthrodesis: severe degenerative changes in the calcaneocuboid joint and/or severe abductus deformity of the forefoot.
* Between the age 18-75

Exclusion Criteria:

* Acute or chronic infection.
* Poor vascular status of the lower leg (relative contraindication for double arthrodesis through a single medial approach).
* Women that are pregnant.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be identified in the clinic by an attending orthopaedic foot and ankle surgeon or his physician assistant based on clinical exam and radiographic findings. Patients of all racial, religious, and cultural backgrounds will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-10-07 (Actual); Primary Completion 2024-01-29 (Actual); Study Completion 2024-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark E. Easley, MD, Principal Investigator — Duke Health
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be available. The results will be statistically analyzed as a whole.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two participants withdrew prior to surgery.
Period: Overall Study
Arm/Group | Aptus CCS 5.0 or/and 7.0 Screws
Started | 48
Completed | 24
Not Completed | 24
Not completed — Lost to Follow-up | 9
Not completed — Withdrawal by Subject | 15

BASELINE CHARACTERISTICS:
Arm/Group | Aptus CCS 5.0 or/and 7.0 Screws
Number analyzed (Participants) | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (15.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 48
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 41
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 48

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Intraoperative Complications
Description: All intraoperative complications including injury of neurovascular structures and/or tendons will be prospectively documented. All intraoperative technical difficulties (for example, breakage of the screw) will be prospectively documented.
Time Frame: At time of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Aptus CCS 5.0 or/and 7.0 Screws
Number analyzed (Participants) | 48
Participants | 0

2. Primary Outcome: Number of Participants With Perioperative Complications
Description: All perioperative complications including wound healing problems and/or superficial/deep infection and/or deep vein thrombosis will be prospectively documented.
Time Frame: Up to 2 years post-operative
Measure: Count of Participants; unit: Participants
Arm/Group | Aptus CCS 5.0 or/and 7.0 Screws
Number analyzed (Participants) | 48
Participants | 28

3. Primary Outcome: Number of Participants With Delayed Osseous Union or Non-union
Description: Independent radiologist will measure fusion of standard of care radiographs and CT scan
Time Frame: Up to 2 years post-operative
Measure: Count of Participants; unit: Participants
Arm/Group | Aptus CCS 5.0 or/and 7.0 Screws
Number analyzed (Participants) | 48
Participants | 4

4. Primary Outcome: Number of Participants With Fixation of a Double or Triple Arthrodesis Neutral Hindfoot Alignment
Description: An independent radiologist will measure fusion of the double, triple, or subtalar fusion by reviewing the standard of care radiographs and CT scan and measuring the rate of fusion using the bridging of the trabecular bone.
Time Frame: Up to 2 years post-operative
Population: Data not collected due to infeasibility.
Arm/Group | Aptus CCS 5.0 or/and 7.0 Screws
Number analyzed (Participants) | 0

5. Primary Outcome: Pain Following Double or Triple Arthrodesis as Measured by a Visual Analogue Scale (VAS)
Description: The VAS ranges from 0 (no pain) to 10 (maximal pain).
Time Frame: Baseline (pre-operative), 3 months, 6 months, 1 year, and 2 years post-operative
Population: Participants with data collected at each timepoint. Two participants withdrew prior to surgery, but had baseline data collected.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aptus CCS 5.0 or/and 7.0 Screws
Number analyzed (Participants) | 50
score on a scale
  Baseline | 6.56 (2.65)
  3 months: number analyzed (Participants) | 40
  3 months | 2.73 (2.60)
  6 months: number analyzed (Participants) | 36
  6 months | 2.34 (2.40)
  1 year: number analyzed (Participants) | 29
  1 year | 2.05 (2.58)
  2 years: number analyzed (Participants) | 23
  2 years | 2.47 (2.45)

6. Primary Outcome: Functional Status Following Double or Triple Arthrodesis as Measured by the American Orthopaedic Foot and Ankle Society (AOFAS) Hindfoot Score
Description: The final score is the sum of the points across all 9 questions with a total score range of 0 to 28. A higher score indicates greater functionality.
Time Frame: Baseline (pre-operative), 6 weeks, 3 months, 6 months, 1 year, and 2 years post-operative
Population: Participants with data collected at each timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aptus CCS 5.0 or/and 7.0 Screws
Number analyzed (Participants) | 46
score on a scale
  Baseline | 18.74 (3.42)
  3 months: number analyzed (Participants) | 28
  3 months | 17.60 (2.30)
  6 months: number analyzed (Participants) | 34
  6 months | 15.38 (2.64)
  1 year: number analyzed (Participants) | 23
  1 year | 13.65 (2.67)
  2 years: number analyzed (Participants) | 14
  2 years | 14.71 (2.20)

7. Primary Outcome: Functional Status Following Double or Triple Arthrodesis as Measured by the Foot & Ankle Disability Index (FADI) Score
Description: The FADI has a total score range of 0 to 104, where a higher score indicates greater functionality.
Time Frame: Baseline (pre-operative), 6 weeks, 3 months, 6 months, 1 year, and 2 years post-operative
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aptus CCS 5.0 or/and 7.0 Screws
Number analyzed (Participants) | 50
score on a scale
  Baseline | 49.02 (16.87)
  3 months: number analyzed (Participants) | 39
  3 months | 47.00 (24.30)
  6 months: number analyzed (Participants) | 36
  6 months | 70.67 (15.81)
  1 year: number analyzed (Participants) | 29
  1 year | 75.76 (19.74)
  2 years: number analyzed (Participants) | 25
  2 years | 78.44 (18.23)

8. Primary Outcome: Number of Participants With Secondary Surgical Procedures for Any Reason Including Hardware Removal
Description: All postoperative complications requiring any secondary surgical procedures including hardware removal will be prospectively documented.
Time Frame: Up to 2 years post-operative
Measure: Count of Participants; unit: Participants
Arm/Group | Aptus CCS 5.0 or/and 7.0 Screws
Number analyzed (Participants) | 48
Participants | 5

ADVERSE EVENTS:
Time Frame: Up to 2 years post-operative
Arm/Group | Aptus CCS 5.0 or/and 7.0 Screws
All-Cause Mortality (participants affected / at risk) | 2/48
Serious Adverse Events (participants affected / at risk) | 8/48
Other Adverse Events (participants affected / at risk) | 26/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aptus CCS 5.0 or/and 7.0 Screws (N=48)
Implant failure (Musculoskeletal and connective tissue disorders) | 3
Deep vein thrombosis (Musculoskeletal and connective tissue disorders) | 1
Hardware Removal (Musculoskeletal and connective tissue disorders) | 5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aptus CCS 5.0 or/and 7.0 Screws (N=48)
Wound Breakdown (Musculoskeletal and connective tissue disorders) | 1
Swelling (Musculoskeletal and connective tissue disorders) | 14
Pain (Musculoskeletal and connective tissue disorders) | 9
Others (Musculoskeletal and connective tissue disorders) | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-31): https://cdn.clinicaltrials.gov/large-docs/38/NCT02619838/Prot_SAP_000.pdf